CLINICAL TRIAL: NCT04461041
Title: Empagliflozin and Cardiac Remodelling in People Without Diabetes
Acronym: EMPA-HEART 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Medical and Surgical Knowledge Translation Research Group (Other); Boehringer Ingelheim (Industry); Applied Health Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1245-0206
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cardiovascular Diseases; Left Ventricular Hypertrophy
Keywords: Cardiovascular disease; Cardiac Magnetic Resonance Imaging; Sodium-Glucose Transporter 2 Inhibitors
MeSH Terms: conditions — Cardiovascular Diseases; Hypertrophy, Left Ventricular | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Active Comparator): Single 10 mg tablet, administered orally once daily for 6 months
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Single 10 mg tablet, administered orally once daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Single oral tablet
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — Placebo tablet manufactured to mimic empagliflozin 10 mg tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of empagliflozin on cardiac structure, function and circulating biomarkers in patients with cardiovascular risk factors, but without diabetes. Empagliflozin is an antihyperglycemic agent approved by Health Canada and the FDA for the treatment of type 2 diabetes. Previous post-marketing clinical trials demonstrated a reduction in cardiovascular deaths and heart failure in patients with type 2 diabetes treated with empagliflozin. In the first EMPA-HEART trial, we demonstrated that empagliflozin reduces cardiac mass in patients with type 2 diabetes, as seen through cardiac magnetic resonance imaging (cMRI). Therefore, the aim of this study, EMPA-HEART 2, is to determine whether empagliflozin can similarly impact cardiac structure in patients without diabetes, but with various cardiovascular risk factors.

DETAILED DESCRIPTION:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors (empagliflozin, canagliflozin and dapagliflozin) are approved medications to improve glycemic control in adult patients with type 2 diabetes. When added to current standard-of-care diabetes treatment, SGLT2 inhibitors are associated with clinically meaningful reductions in major adverse cardiovascular events, reduced rates of hospitalization for heart failure and a decrease in major adverse kidney outcomes. Importantly, these benefits were observed consistently in people with and without type 2 diabetes and across all levels of baseline glycemic control. These data point towards a glucose-independent, cardioprotective effect of SGLT2 inhibition. How SGLT2 inhibition might reduce cardiac outcomes in people without diabetes remains unclear, and this is the specific objective of EMPA-HEART 2.

The study drug, empagliflozin (marketed as Jardiance), belongs to a class of medications that lowers blood glucose (sugar) by preventing glucose from entering back into blood circulation and ensures it is eliminated in urine. Empagliflozin is approved by the FDA and Health Canada for the treatment of type 2 diabetes.

This is a double-blind, randomized, placebo-controlled, parallel-group study of empagliflozin vs. placebo in patients without diabetes but with various cardiovascular risk factors. The purpose is to determine the effects of empagliflozin on cardiac structure by using cMRI. Patients who have given informed consent will undergo a baseline cMRI and will then be randomly assigned in a 1:1 basis to either empagliflozin 10 mg once daily or matching placebo. An end of study cMRI will be performed at 26 weeks (6 months after starting the study drug).

The study subjects will be followed for 6 months. The patients will be assessed using cMRI, which is considered the "gold standard" for measuring left ventricular (LV) volume, mass, and ejection fraction. The investigators will assess changes from baseline in LV mass, LV end-diastolic volume, end-systolic volume, LV ejection fraction, LV diastolic and systolic function, and LV wall stress via cMRI in enrolled patients treated with empagliflozin compared to those who receive placebo. Additionally, changes from baseline in blood pressure, hematocrit, and biomarkers involved in the pathophysiology of heart failure, namely NT-proBNP, will be evaluated at 6 months.

Study assessments and potential adverse events reporting will be undertaken at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Female Not of childbearing potential and male subjects ≥ 18 and ≤ 85 years of age (Women Not of childbearing potential are females who are permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause or ≥6 weeks post-surgical bilateral oophorectomy prior to Screening.)
2. ≥1 of the major criteria or ≥2 of the minor criteria below:

   Major criteria
   * Increased LVMi of ≥96 g/m2 for women and ≥116 g/m2 for men (as calculated by echocardiogram); or LVMi ≥81 g/m2 for women and ≥85 g/m2 for men (as calculated by cMRI)
   * ECG evidence of LV hypertrophy (as per the Sokolow-Lyon criteria)
   * Structural heart disease defined as interventricular septal thickness or posterior wall thickness at end-diastole of ≥11 mm (as measured by 2D echocardiography or cMRI)
   * Persistent hypertension (defined as office blood pressure ≥140/90 mmHg) despite being on ≥3 antihypertensive medications

   Minor criteria
   * Prior history of a myocardial infarction (≥3 months ago)
   * eGFR ≥30 and ≤60 mL/min/1.73 m2 (as measured by the CKD-EPI formula)
   * Body mass index (BMI) ≥27 kg/m2
3. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures

Exclusion Criteria:

1. Female subjects who are pregnant, lactating or of childbearing potential, or are pre-menopausal
2. Known type 1 or type 2 diabetes
3. Hemoglobin A1C (A1C) ≥6.5%
4. eGFR <30 mL/min/1.73m2
5. Known history of severe liver disease (e.g. Child Pugh Class B or C)
6. Known history of severe symptomatic untreated anemia in the last 3 months (e.g. hemoglobin < 90 g/L)
7. History of ketoacidosis, or increased chance of developing diabetic ketoacidosis (DKA) e.g. patients who suffer from excessive vomiting, diarrhea, or sweating; subjects who are on a very low carbohydrate diet; or subjects who drink a lot of alcohol.
8. Systolic blood pressure <95mmHg (as measured at the office/clinic visit)
9. Subjects in whom coronary revascularization by either percutaneous coronary intervention or bypass surgery is being contemplated within the next 6 months, or who have undergone coronary revascularization in the prior 3 months
10. Significant allergy or known intolerance to SGLT2is or any ingredient in the formulations
11. Subjects currently experiencing any clinically significant or unstable medical condition that in the opinion of the investigator might limit their ability to complete the study, or to comply with the requirements of the protocol, including: dermatologic disease, hematological disease, pulmonary disease, hepatic disease, gastrointestinal disease, genitourinary disease, endocrine disease, neurological disease, and psychiatric disease
12. Any malignancy not considered cured (except basal cell carcinoma of the skin). A subject is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening
13. Subjects who have participated in other interventional studies which may affect any of the primary or secondary outcomes of the study within 30 days of the screening visit
14. Contraindications or inability to undergo magnetic resonance imaging such as severe obesity (e.g. weight >500 lbs) or the presence of metallic fragments, clips, or devices
15. Known history of infiltrative cardiomyopathy such as cardiac amyloidosis or cardiac sarcoidosis
16. Severe aortic stenosis
17. Severe aortic regurgitation
18. Severe mitral stenosis
19. Severe mitral regurgitation
20. Low voltage on ECG limb leads defined by the amplitude of the QRS complex in each limb lead ≤0.5 mV

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Left Ventricular (LV) mass | 6 months
  Change in Left Ventricular (LV) mass (indexed to body surface area (BSA)) at 6 months. This will be measured using CMRI.

SECONDARY OUTCOMES:
LV end-diastolic volume | 6 months
  Change in LV end-diastolic volume (indexed to BSA) at 6 months. This will be measured using CMRI.
LV end-systolic volume | 6 months
  Change in LV end-systolic volume (indexed to BSA) at 6 months. This will be measured using CMRI.
Left Ventricular Ejection Fraction (LVEF) | 6 months
  Change in LVEF at 6 months. This will be measured using CMRI.
LV wall stress | 6 months
  Change in LV wall stress at 6 months. This will be measured using CMRI.
LV systolic function | 6 months
  Change in LV systolic function at 6 months. This will be measured using CMRI.
LV diastolic function | 6 months
  Change in LV diastolic function at 6 months. This will be measured using CMRI.
NT-proBNP | 6 months
  Change in circulating NT-proBNP at 6 months.
Systolic and diastolic blood pressure | 6 months
  Change in systolic and diastolic blood pressure at 6 months.
Hematocrit | 6 months
  Change in hematocrit at 6 months in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD PhD, Principal Investigator — Unity Health Toronto
Locations (4):
- Canada (3):
  - Diagnostic Assessment Centre (AMS Diagnostics), Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - North York Diagnostic and Cardiac Centre, Toronto, Ontario
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Connelly KA, Mazer CD, Puar P, Teoh H, Wang CH, Mason T, Akhavein F, Chang CW, Liu MH, Yang NI, Chen WS, Juan YH, Opingari E, Salyani Y, Barbour W, Pasricha A, Ahmed S, Kosmopoulos A, Verma R, Moroney M, Bakbak E, Krishnaraj A, Bhatt DL, Butler J, Kosiborod MN, Lam CSP, Hess DA, Rizzi Coelho-Filho O, Lafreniere-Roula M, Thorpe KE, Quan A, Leiter LA, Yan AT, Verma S. Empagliflozin and Left Ventricular Remodeling in People Without Diabetes: Primary Results of the EMPA-HEART 2 CardioLink-7 Randomized Clinical Trial. Circulation. 2023 Jan 24;147(4):284-295. doi: 10.1161/CIRCULATIONAHA.122.062769. Epub 2022 Nov 6. PMID 36335517